CLINICAL TRIAL: NCT02348736
Title: Comparative Study Between SensaScope Intuboscope and McGrath Series 5 Videolaryngoscope to Tracheal Intubation: a Prospective Randomised Study
Brief Title: Comparison of SensaScope Intuboscope and McGrath Series 5 for Endotracheal Intubation
Acronym: SensaScope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Marc Kriege,MD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGUM
Record Dates: First submitted 2015-01-12; First posted 2015-01-28 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Airway Morbidity
Keywords: airway; videolaryngoscope
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SensaScope (Experimental): Time for tracheal intubation with the SensaScope
  Interventions: Device: Time for tracheal intubation
- McGrath Series 5 (Experimental): Time for tracheal intubation with the McGrath Series 5
  Interventions: Device: Time for tracheal intubation

INTERVENTIONS:
Device: Time for tracheal intubation — In a randomised trial we measure the time for ventilation by means of endtidale CO2 Curve

SUMMARY:
A randomized controlled prospective study of laryngoscopy and intubation time comparing SensaScope and the McGrath® Series 5 video laryngoscope.

DETAILED DESCRIPTION:
The use of videolaryngoscopy is increasing as a technique for rescue intubation as well as for elective intubation. Current airway management guidelines recommend video-assisted laryngoscopy as a choice for basic airway management. This is a proposed comparison study of a video laryngoscope, use in the daily anesthesia practice, and its likely increased success compared to semi-rigid stylet. An national, mono center, prospective randomized comparative trial (RCT) is proposed testing the superiority of oral tracheal intubation with the McGrath® Series 5 versus SensaScope in adult patients under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years No concurrent participation in another study
* capacity to consent
* Present written informed consent of the research participant
* Elective surgery under general anesthesia

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* emergency patients
* Emergency situations in the context of a Difficult Airway Management
* ASA classification> 3
* situations where the possibility of accumulated gastric contents
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
comparison of different time for tracheal intubation | <2min
  times for tracheal intubation, View of the glottic, experience in anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Negishi Y, Shimada N, Urayama M, Niwa Y, Takeuchi M. [McGRATH MAC Videolaryngoscope: clinical assessment of its performance in 50 surgical patients]. Masui. 2014 Sep;63(9):1025-8. Japanese. PMID 25255665
- [Result] Biro P. The SensaScope- A new hybrid video intubation stylet. Saudi J Anaesth. 2011 Oct;5(4):411-3. doi: 10.4103/1658-354X.87271. PMID 22144929
- [Result] Biro P, Battig U, Henderson J, Seifert B. First clinical experience of tracheal intubation with the SensaScope, a novel steerable semirigid video stylet. Br J Anaesth. 2006 Aug;97(2):255-61. doi: 10.1093/bja/ael135. Epub 2006 Jun 1. PMID 16740606